CLINICAL TRIAL: NCT05865314
Title: Optimised Nutritional Therapy and Early Physiotherapy in Long Term ICU Patients: a Randomized Controlled Study (NutriPhyT Trial)
Brief Title: Optimised Nutritional Therapy and Early Physiotherapy in Long Term ICU Patients (NutriPhyT Trial)
Acronym: NutriPhyT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HEIDEGGER CP (Other)
Responsible Party: Sponsor-Investigator, HEIDEGGER CP, Deputy head physician, Head of the Intensive Care Polyvalent Unit, Division of Intensive Care, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NutriPhyT2022
Record Dates: First submitted 2023-03-23; First posted 2023-05-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; ICU Acquired Weakness; Malnutrition
Keywords: Early nutrition therapy; Early mobilisation; Long stay ICU patient; Physiotherapy
MeSH Terms: conditions — Critical Illness; Malnutrition | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental)
  Interventions: Other: Optimisation of nutrition therapy coupled with early mobilisation
- Control group (Active Comparator)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Optimisation of nutrition therapy coupled with early mobilisation — Optimisation of nutrition therapy coupled with early mobilisation with:
  * Optimisation of nutrition therapy during ICU stay
  * Optimisation of physiotherapy during ICU stay
  * Better communication and closer collaboration between physiotherapy and nutrition teams.
  * Optimisation of continuity of the care.
  Arms: Interventional group
Other: Standard care — Patients will receive nutritional therapy and mobilisation according to local standard procedures.
  Arms: Control group

SUMMARY:
Due to medical advances and quality of care, mortality in adult intensive care units (ICUs) has decreased significantly in recent years, leading to a significant increase in the number of patients with high rehabilitation needs on discharge from the ICU.

A specific management by a multidisciplinary team has been set up since 2017 at the Geneva-ICU for long-stay patients (hospitalised ≥ 7 days).

This study aim to assess whether an optimization of the nutritional therapy coupled with an early mobility during and after the ICU stay allows an improvement in the muscle function at hospital discharge compared to patients receiving the standard care.

DETAILED DESCRIPTION:
Due to medical advances and quality of care, mortality in adult intensive care units (ICUs) has decreased significantly in recent years, leading to a significant increase in the number of patients with high rehabilitation needs on discharge from the ICU. Indeed, these patients are at high risk of complications related to their ICU stay (cognitive impairment, ICU acquired weakness, diaphragm dysfunction, ICU polyneuropathy, post-traumatic stress, malnutrition, etc.). Despite prolonged periods of rehabilitation, there is a significant decrease in functional status and quality of life compared to the previous status of these patient.

A specific management by a multidisciplinary team has been set up since 2017 at the Geneva-ICU for long-stay patients (hospitalised ≥ 7 days) including special attention to weaning from ventilation, nutrition, mobilisation, anxiety, pain, skin condition etc.

The culture of nutritional therapy and early mobilisation is already well established at the Geneva-ICU. However, a comprehensive approach to nutrition and mobilisation during and after the ICU stay could be optimised.

The objective of the study is to determine whether optimization of nutritional therapy combined with early mobilization for patients with long ICU stay will improve muscle function at discharge compared with patients receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

Any patient admitted to the adult ICU :

* ≥18 years old
* On mechanical ventilation with an expected length of stay ≥ 7 days
* Requiring artificial nutrition (enteral and/or parenteral nutrition)

Exclusion Criteria:

Therapeutic withdrawal Pregnant or breastfeeding patients

Neurological disorders with motor deficits:

* New or pre-existing neuromuscular or nervous system disease
* Spinal cord injury Severe polytrauma of the lower limbs (amputation etc.) Non-independent ambulation (including walking aids) before ICU admission

For organizational reasons not allowing follow-up :

* Transfer to another ICU
* Patient living abroad from Switzerland
* Patient living in nursing homes preceding to ICU admission
* Incarcerated patients
* Intellectual/cognitive disabilities or language barrier, limiting ability to follow the instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Walking distance | Hospital discharge or end of the intervention (4 weeks after ICU discharge)
  6 MWT

SECONDARY OUTCOMES:
Walking distance | At ICU discharge (if achievable); 6 months post-ICU stay
  6 MWT
Body composition | At ICU discharge; at hospital discharge or end of the intervention; at 6 months post-ICU stay
  Electrical bio impedance
Body composition | Within the 1st 48 hours post ICU admission, at ICU discharge; at hospital discharge or end of the intervention; at 6 months post-ICU stay
  Peripheral muscle ultrasound
Grip Strength | At ICU discharge; at hospital discharge or end of the intervention; at 6 months post-ICU stay
  Handgrip
Gradation of muscle function | At ICU discharge; at hospital discharge or end of the intervention; at 6 months post-ICU stay
  MRC
Physical functionality | At ICU discharge; at hospital discharge or end of the intervention; at 6 months post-ICU stay
  PFIT & SPPB
Weight difference | At ICU admission, at ICU discharge; at hospital discharge or end of the intervention; at 6 months post-ICU stay
  Comparison between weight at ICU admission, at hospital discharge and at 6 months post-ICU stay
Appetite | At ICU discharge; at hospital discharge or end of the intervention; at 6 months post-ICU stay
  10-point survey scale
Food intake estimation | At 6 months post-ICU stay
  3 days food diary
Quality of life (SF-12) | At 6 months post-ICU stay
  SF-12
Return to work/activity preceding to the event | At 6 months post-ICU stay
  Collected during the 6 month post-ICU stay consultation
Length of ICU and hospital stay | At ICU and hospital discharge
  Collected in the patient form
Duration of mechanical ventilation | At ICU discharge
  Collected in the patient form

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Heidegger, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Service of Intensive Care, Geneva University Hospital,, Geneva, Canton of Geneva, Switzerland